CLINICAL TRIAL: NCT03326791
Title: Acetylsalicylic Acid as Secondary Prevention in Colorectal Cancer
Brief Title: Aspirin in Colorectal Cancer Liver Metastases
Acronym: ASAC
Status: Active, not recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Collaborators: Norwegian Cancer Society (Other); The Research Council of Norway (Other); Klinbeforsk (Other)
Responsible Party: Principal Investigator, Sheraz Yaqub, MD PhD, Coordinating Investigator, Oslo University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2014/2217
Record Dates: First submitted 2017-10-02; First posted 2017-10-31 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Colorectal Cancer Liver Metastases; Colorectal Cancer; Liver Metastases
Keywords: Acetylsalicylic acid; Aspirin; Trombyl; Secondary prevention
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Aspirin

STUDY DESIGN:
Intervention Model Description: Multi-centre, double-blinded, randomized, placebo-controlled clinical intervention trial.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Eligible patients will be allocated in a 1:1 ratio using a computer randomization procedure stratified by centre. The randomization will be blocked within each stratum.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention group (Experimental): Acetylsalicylic acid 160 mg once daily until recurrent disease or a total period of 3 years.
  Interventions: Drug: Acetylsalicylic acid
- Control group (Placebo Comparator): Placebo Oral Tablet once daily until recurrent disease or a total period of 3 years.
  Interventions: Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: Acetylsalicylic acid — Trombyl 160 mg once daily
  Other Names: Trombyl; Aspirin
  Arms: Intervention group
Drug: Placebo Oral Tablet — Placebo one tablet daily
  Arms: Control group

SUMMARY:
The ASAC trial is a Scandinavian, multi-center, double-blinded, randomized, placebo-controlled study to determine whether adjuvant treatment with low-dose acetylsalicylic acid (ASA) can improve disease free survival in patients treated with resection for colorectal cancer liver metastases (CRCLM).

Several studies have shown beneficial effect of ASA on primary prevention of CRC and the investigators group and others have shown a potential association of ASA also taken after the diagnosis on CRC survival in registry-based studies (secondary prevention). Up to 800 patients operated for CRCLM will be randomized to Arm#1 ASA 160 mg once daily or Arm#2 Placebo for a period of 3 years or till disease recurrence. The patients will be treated and followed up according to standard of care and the National Guidelines.

The ASAC trial will be the first clinical interventional trial to assess the beneficial role of ASA in recurrence of CRC liver metastases and survival. ASA is an inexpensive, well tolerated, and easily accessible drug that will be highly potential as adjuvant drug in secondary prevention of CRC liver metastases if the study shows a beneficial effect. This trial will also investigate the effect of ASA as adjuvant treatment on Health-related Quality of Life and the cost-effectiveness.

ELIGIBILITY:
Inclusion Criteria:

* First time CRCLM (synchronous or metachronous).
* Recurrence of CRCLM (not previously included in this trial).
* In synchronous CRCLM and "Liver first" approach, the primary tumor must be resected within 6 weeks after the liver
* Macroscopic (surgical) free resection margins (R0 or R1 resection).
* Must be ambulatory with a performance status Eastern Cooperative Oncology Group (ECOG) 0-2.
* Must be at least 18 years of age.
* Signed informed consent and expected cooperation of the patients for the treatment and follow up must be obtained and documented according to International Conference on Harmonization - Good Clinical Practice (ICH GCP), and national/local regulations.

Exclusion Criteria:

* Concomitant use of ASA or other anticoagulants or platelet inhibitors such as warfarin or clopidogrel.
* Ongoing regular use of corticosteroids or NSAIDs.
* Inherited or acquired coagulopathy (haemophilia).
* Blood platelets (thrombocytes) < 100 x 10^9/L.
* Severe heart failure (classified as New York Heart Association (NYHA) class >III)
* Severe kidney failure >Stage 3b
* CRCLM previously treated with radiofrequency or microwave ablation technique
* Pregnancy or breastfeeding. For women in childbearing age there will be pregnancy test at monthly intervals (urine human chorionic gonadotropin (HCG) pregnancy tests (for home testing) will be given to the patients for monthly tests and the patient will self-report the results at each control). Furthermore, highly effective contraceptives will be required.
* Childbearing potential without proper contraceptive measures such as oral contraceptives, other hormonal contraceptives (vaginal products, skin patches, or implanted or injectable products), or mechanical products such as an intrauterine device to avoid pregnancy for the entire study period.
* Liver cirrhosis with a Child-Pugh score >B7.
* Alcoholism.
* Contraindication listed on the Summary of Product Characteristics (SmPC) of Trombyl: Hypersensitivity/allergies to ASA, Thrombocytopenia, Previous severe gastrointestinal haemorrhage/peptic ulcer due to ASA/NSAID, Active peptic ulcer, Haemophilia, Liver cirrhosis, Severe congestive heart failure.
* Need to use concomitant medications contraindicated according to SmPC of Trombyl.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 466 (Actual)
Dates: Start 2017-12-15 (Actual); Primary Completion 2022-02-01 (Actual); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Disease Free Survival (DFS) after three years treatment | 3 years
  DFS three years after initiation of treatment with ASA or Placebo after resection of liver metastases.

SECONDARY OUTCOMES:
Time to recurrence (TTR) of disease after randomization | 3 years
  Time to recurrence of liver metastases three years after start of treatment.
Overall survival (OS) three years after treatment start | 3 years
  OS at three years after initiation of treatment with ASA or Placebo
Health-related Quality of Life with 36-item Short Form Health Survey (SF-36) | 3 years
  SF-36 has been proven useful in monitoring population health, estimating the burdens of different diseases, monitoring outcome in clinical practice, and evaluating medical treatment effects. Health-related Quality of Life (HR-QoL) will be assessed with SF-36.
Health-related Quality of Life with EuroQoL 5 Dimensions (EQ-5D) | 3 years
  The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. The EQ VAS records the patient's self-rated health on a vertical visual analogue scale. This will be used as a quantitative measure of health outcome that reflects the patient's own judgement. The scores on these five dimensions will be presented as a health profile. Health-related Quality of Life (HR-QoL) will be assessed with EuroQoL 5 Dimensions (EQ-5D).
ASA in CRC and Cost-Effectiveness Analyses I | 3 years
  Changes in HR-QoL will be used in calculation of the quality-adjusted life-year (QALY), a key outcome used in economic evaluations to compare treatments.
ASA in CRC and Cost-Effectiveness Analyses II | 3 years
  Cost-effectiveness measured from a health care perspective by assessing the use of Health care provider in primary and specialized medicine.
ASA in CRC and Cost-Effectiveness Analyses III | 3 years
  Cost-effectiveness measured from a societal perspective by assessing records in Statistics Norway (SSB).

CONTACTS AND LOCATIONS:
Overall Officials: Kjetil Taskèn, MD PhD, Principal Investigator — University of Oslo; Sheraz Yaqub, MD PhD, Principal Investigator — Oslo University Hospital
Locations (14):
- Denmark (3):
  - Aarhus University Hospital, Aarhus, Aarhus
  - Rigshospitalet, Copenhagen, Copenhagen, Copenhagen
  - Odense University Hospital, Odense
- Norway (5):
  - Haukeland University Hospital, Bergen, Bergen
  - Oslo University Hospital, Oslo, Oslo County
  - Stavanger University Hospital, Stavanger, Stavanger
  - University Hospital of North-Norway, Tromsø, Tromsø
  - St Olavs Hospital, Trondheim, Trondheim
- Sweden (6):
  - Sahlgranska University Hospital, Gothenburg, Gothenburg
  - Linköping University Hospital, Linköping, Linköping
  - Skåne University Hospital Lund, Lund, Lund
  - Karolinska University Hospital, Stockholm, Stockholm County
  - Uppsala University Hospital, Uppsala, Uppsala County
  - University Hospital of Umeå, Umeå

REFERENCES:
- [Derived] Yaqub S, Bjornbeth BA, Angelsen JH, Fristrup CW, Gronbech JE, Hemmingsson O, Isaksson B, Juel IS, Larsen PN, Lindell G, Mortensen FV, Mortensen KE, Rizell M, Sandstrom P, Sandvik OM, Sparrelid E, Taflin H, Tasken K; ASAC study group. Aspirin as secondary prevention in colorectal cancer liver metastasis (ASAC trial): study protocol for a multicentre randomized placebo-controlled trial. Trials. 2021 Sep 20;22(1):642. doi: 10.1186/s13063-021-05587-w. PMID 34544470
- See also: Website — http://www.asac.no/
- See also: Related Info — https://kliniskestudier.helsenorge.no/tykktarmskreft-kan-acetylsalisylsyre-hindre-tilbakefall-av-spredning